CLINICAL TRIAL: NCT07354347
Title: Optimal ATP Settings in the VT Zone for New Implantable Cardioverter Defibrillator (ICD) Implantation (DAN-ATP)
Brief Title: Optimal Settings for Anti Tachycardia Pacing (ATP) on ICD
Acronym: DAN-ATP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Bo Gregers Winkel, Chief Physician, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAN-ATP; 2501444 (Other: VMK)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Heart Disease; Implantable Cardioverter Defibrillator (ICD); Heart Rhythm Disorders; Ventricular Tachyarrhythmias
Keywords: Heart failure; ICD; ATP; Anti Takykardi Pacing; Implantable Cardioverter Defibrillator; cluster randomisation; heart rhythm disorder; ventricular tachyarrhythmias; VT
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Tachycardia, Ventricular; Heart Failure | interventions — Architectural Accessibility

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic, two-group, cluster randomized trial. With clusters of time periods of 4-month duration at all sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst (Experimental)
  Interventions: Other: Burst
- Ramp (Experimental)
  Interventions: Other: Ramp

INTERVENTIONS:
Other: Burst — ATP with 4 burst
  Arms: Burst
Other: Ramp — ATP with 1 Burst + 3 Ramp
  Arms: Ramp

SUMMARY:
This is a pragmatic, two-group, cluster randomized trial designed to compare strategies for the Anti Tachycardia Pacing (ATP)-setting in the ventricular tachyarrhythmias (VT) zone when implanting a new implantable cardioverter defibrillator (ICD) in patients with heart disease in hospitals in Denmark.

The strategies are: "Burst" or "Ramp" after 1. ATP (which is always burst) in VT zone. VT zone is defined between 180-249 (up to 269 in special cases) heartbeats per minute.

The ICD will give either:

Burst: The ICD is programmed to give ATP with 4 bursts. Or Ramp: The ICD is programmed to give ATP with 1 burst and 3 ramps.

The participating hospitals will be assigned to one of two intervention strategies for periods of 4-months. The given intervention will follow the patient/ICD throughout the life time of the ICD, but with the possibility to reprogram at any time (intention to treat).

It is calculated that the study needs a total of 398 events (second to fourth ATP), which is estimated to require 3980 implanted ICDs. The participants will be followed until the end of the ICD life, which is estimated to be around 10 years.

ELIGIBILITY:
Inclusion Criteria:

- ICD implantation for primary or secondary prophylactic indication

Exclusion Criteria:

* None
* Patients can actively opt out of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3980 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2041-07-31 (Estimated); Study Completion 2041-07-31 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia cessation | The lifetime of the ICD, estimated 10 years
  The ability of the given ATP protocol to stop the ventricular arrhythmia

SECONDARY OUTCOMES:
Defibrillation | The lifetime of the ICD, estimated 10 years
  Arrhythmia accelerates resulting in defibrillation/shock therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The Heart Center, Rigshospitalet, Copenhagen, Dr., Denmark

IPD SHARING:
Plan to Share IPD: No
The data are considered sensitive personal data.